CLINICAL TRIAL: NCT04309175
Title: Effect of Long-term Atrial Pacing on Central Blood Pressure in Permanently Paced Sick Sinus Syndrome Patients With Primary Arterial Hypertension
Brief Title: Long-term Atrial Pacing and Central Blood Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tartu University Hospital (Other)
Collaborators: North Estonia Medical Centre (Other)
Responsible Party: Principal Investigator, Tuuli Teeäär, cardiologist, Tartu University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 299/T-22
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Blood Pressure
Keywords: central blood pressure; sick sinus syndrome; pacemaker; hypertension; sinus node dysfunction
MeSH Terms: conditions — Sick Sinus Syndrome; Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Slow-Fast (Experimental)
  Interventions: Device: base rate programming of a permanent cardiac pacemaker
- Fast-Slow (Experimental)
  Interventions: Device: base rate programming of a permanent cardiac pacemaker

INTERVENTIONS:
Device: base rate programming of a permanent cardiac pacemaker — Base rate of a subject's pacemaker is set to a slower, and after wash-out, to a faster pacing rate (Slow-Fast Arm) or to a faster, and after wash-out, to a slower pacing rate (Fast-Slow Arm)

SUMMARY:
This is a randomized controlled single-centre clinical trial with a cross-over design to compare non-invasively evaluated central blood pressure and related parametres in sick sinus syndrome patients with hypertension who are paced long-term at a slower vs faster heart rate

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years
* sick sinus syndrome
* permanent cardiac pacemaker with right atrial and right ventricular leads
* at least 3 months from implantation
* sinus rhythm
* percentage of atrial pacing at or above 80% since last interrogation
* percentage of ventricular pacing at or below 3% since last interrogation
* primary arterial hypertension
* antihypertensive drug treatment
* mean office brachial blood pressure below 140/90 mmHg
* mean home brachial blood pressure below 135/85 mmHg
* ability to understand and follow study protocol
* signed informed consent form

Exclusion Criteria:

* inclusion criteria not fulfilled
* violation of study protocol by subject, investigator or third part
* high quality central hemodynamic measurements cannot be perfomed
* inter-arm difference in brachial systolic blood pressure 15 mmHg or above
* intrinsic QRS complex 130 ms or above
* more than three antihypertensive agents in use
* treatment with digoxin or agents from Vaughan-Williams classes Ic, III või IV
* frequent high atrial rate episodes
* coronary artery disease
* secondary hypertension
* resistant hypertension
* orthostatic hypotension
* heart failure with decreased or preserved left ventricular ejection fraction
* implantable cardioverter-defibrillator or cardiac resynchronization therapy
* significant valvular heart disease
* significant congenital heart disease
* body mass index ≥35 kg/m2
* type I diabetes
* type II diabetes with cardiovascular complications or on insulin therapy
* other significant endocrine disease
* history of cerebrovascular attack
* carotid artery disease
* lower extremity arterial disease
* severe chronic obstructive pulmonary disease
* severe asthma
* severe sleep apnea
* interstitial pulmonary disease
* inhaled beta adrenergic agonist therapy
* active cancer treatment
* central nervous system degenerative disease
* systemic connective tissue disease
* abnormal TSH at present
* glomerular filtration rate ≤30 ml/min/m2
* hemoglobin <100 g/L (female), <110 g/L (male)
* hepatic dysfunction
* alcohol abuse
* pregnancy or breastfeeding
* no health insurance provided by Estonian Health Insurance Fund
* withdrawal of informed consent
* loss of contact with a subject during study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
systolic blood pressure amplification change | two months

IPD SHARING:
Plan to Share IPD: Undecided